CLINICAL TRIAL: NCT01893853
Title: Fluid Balance During Exercise in the Heat With Water, Flavored Placebo, or a Carbohydrate-electrolyte Beverage Intake (The APEX Study)
Acronym: APEX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: PBRC 12038
Record Dates: First submitted 2013-06-17; First posted 2013-07-09 (Estimated); Last update posted 2022-09-15 (Actual); Status verified 2022-09

CONDITIONS: Dehydration
Keywords: dehydration; fluid balance; exercise; heat; body weight; performance
MeSH Terms: conditions — Dehydration; Motor Activity; Body Weight

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Water (Other): Electrolyte- and mineral-free water with exercise intervention
  Interventions: Other: Exercise Intervention
- Placebo (Placebo Comparator): Calorie- and electrolyte-free, sweetened flavored water with exercise intervention
  Interventions: Other: Exercise Intervention
- Carbohydrate-electrolyte beverage (Experimental): Commercially-available flavored beverage carbohydrate-electrolyte beverage with Exercise Intervention
  Interventions: Other: Exercise Intervention

INTERVENTIONS:
Other: Exercise Intervention — Exercise intervention trials will consist of a steady-state bout of exercise at ~70% VO2peak and a timed performance test on a cycle ergometer in a heated environment.

SUMMARY:
The purpose of the APEX study is to determine whether carbohydrate-electrolyte beverage intake promotes fluid balance during exercise in the heat compared with water or placebo intake.

DETAILED DESCRIPTION:
Exercise in the heat has large effects on cardiovascular strain, the ability to regulate core body temperature, and performance because of an increase in the reliance on body fluid distribution to the skin to maintain adequate sweat rates and heat dissipation. Carbohydrate-electrolyte beverage intake during exercise in the heat may improve fluid balance and subsequent physical performance.

The participants will be assigned each arm in a randomized, counterbalanced, cross-over fashion separated by at least 2 weeks. Participants will be placed in a heated environment for the duration of the exercise intervention.

ELIGIBILITY:
Inclusion Criteria:

* Males aged 18-35 years
* Healthy (No uncontrolled disease)

Exclusion Criteria:

* No medications that influence fluid balance
* No uncontrolled disease

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Fluid Balance | 120 minutes
  Fluid balance will be determined by change in body weight during the 120 minutes steady-state exercise bout in the heat.

SECONDARY OUTCOMES:
Rate of fluid uptake in the GI tract | 30 minutes
  Fluid uptake in the GI tract be assessed by D20 accumulation in the plasma.
Amount of carbohydrate oxidized | 120 minutes
  Carbohydrate oxidation rates will be assessed by indirect calorimetry.
Cardiovascular responses | 120 minutes
  Heart rate and blood pressure will be assessed during exercise.
Thermoregulatory responses | 120 minutes
  Body temperatures will be assessed during exercise.
Physical Performance | 30 minutes
  Performance during the timed exercise trial will be improved with carbohydrate-electrolyte beverage intake compared with water and placebo intake.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy S Church, MD, MPH, PhD, Principal Investigator — Pennington Biomedical Research Center; Neil M Johannsen, PhD, Study Chair — Louisiana State University-Department of Kinesiology; Ronald B Monce, PA-c, Study Chair — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

REFERENCES:
- [Background] Latzka WA, Sawka MN, Montain SJ, Skrinar GS, Fielding RA, Matott RP, Pandolf KB. Hyperhydration: thermoregulatory effects during compensable exercise-heat stress. J Appl Physiol (1985). 1997 Sep;83(3):860-6. doi: 10.1152/jappl.1997.83.3.860. PMID 9292474
- [Background] Latzka WA, Sawka MN, Montain SJ, Skrinar GS, Fielding RA, Matott RP, Pandolf KB. Hyperhydration: tolerance and cardiovascular effects during uncompensable exercise-heat stress. J Appl Physiol (1985). 1998 Jun;84(6):1858-64. doi: 10.1152/jappl.1998.84.6.1858. PMID 9609777
- [Background] Armstrong LE, Costill DL, Fink WJ. Influence of diuretic-induced dehydration on competitive running performance. Med Sci Sports Exerc. 1985 Aug;17(4):456-61. doi: 10.1249/00005768-198508000-00009. PMID 4033401
- [Background] Cheuvront SN, Carter R 3rd, Castellani JW, Sawka MN. Hypohydration impairs endurance exercise performance in temperate but not cold air. J Appl Physiol (1985). 2005 Nov;99(5):1972-6. doi: 10.1152/japplphysiol.00329.2005. Epub 2005 Jul 14. PMID 16024524
- [Background] Greenleaf JE, Sargent F 2nd. Voluntary dehydration in man. J Appl Physiol. 1965 Jul;20(4):719-24. doi: 10.1152/jappl.1965.20.4.719. No abstract available. PMID 5838723
- [Background] Hubbard RW, Sandick BL, Matthew WT, Francesconi RP, Sampson JB, Durkot MJ, Maller O, Engell DB. Voluntary dehydration and alliesthesia for water. J Appl Physiol Respir Environ Exerc Physiol. 1984 Sep;57(3):868-73. doi: 10.1152/jappl.1984.57.3.868. PMID 6490470
- [Background] Hamilton MT, Gonzalez-Alonso J, Montain SJ, Coyle EF. Fluid replacement and glucose infusion during exercise prevent cardiovascular drift. J Appl Physiol (1985). 1991 Sep;71(3):871-7. doi: 10.1152/jappl.1991.71.3.871. PMID 1757323
- [Background] Nose H, Mack GW, Shi XR, Nadel ER. Role of osmolality and plasma volume during rehydration in humans. J Appl Physiol (1985). 1988 Jul;65(1):325-31. doi: 10.1152/jappl.1988.65.1.325. PMID 3403476
- [Background] Nose H, Mack GW, Shi XR, Nadel ER. Involvement of sodium retention hormones during rehydration in humans. J Appl Physiol (1985). 1988 Jul;65(1):332-6. doi: 10.1152/jappl.1988.65.1.332. PMID 3042742
- [Background] Wilk B, Bar-Or O. Effect of drink flavor and NaCL on voluntary drinking and hydration in boys exercising in the heat. J Appl Physiol (1985). 1996 Apr;80(4):1112-7. doi: 10.1152/jappl.1996.80.4.1112. PMID 8926234
- [Background] Rivera-Brown AM, Gutierrez R, Gutierrez JC, Frontera WR, Bar-Or O. Drink composition, voluntary drinking, and fluid balance in exercising, trained, heat-acclimatized boys. J Appl Physiol (1985). 1999 Jan;86(1):78-84. doi: 10.1152/jappl.1999.86.1.78. PMID 9887116
- [Background] Wemple RD, Morocco TS, Mack GW. Influence of sodium replacement on fluid ingestion following exercise-induced dehydration. Int J Sport Nutr. 1997 Jun;7(2):104-16. doi: 10.1123/ijsn.7.2.104. PMID 9189781
- [Background] Szlyk PC, Sils IV, Francesconi RP, Hubbard RW, Armstrong LE. Effects of water temperature and flavoring on voluntary dehydration in men. Physiol Behav. 1989 Mar;45(3):639-47. doi: 10.1016/0031-9384(89)90085-1. PMID 2756057
- [Background] Vrijens DM, Rehrer NJ. Sodium-free fluid ingestion decreases plasma sodium during exercise in the heat. J Appl Physiol (1985). 1999 Jun;86(6):1847-51. doi: 10.1152/jappl.1999.86.6.1847. PMID 10368348
- [Background] American College of Sports Medicine; Sawka MN, Burke LM, Eichner ER, Maughan RJ, Montain SJ, Stachenfeld NS. American College of Sports Medicine position stand. Exercise and fluid replacement. Med Sci Sports Exerc. 2007 Feb;39(2):377-90. doi: 10.1249/mss.0b013e31802ca597. PMID 17277604
- [Background] Mitchell JW, Nadel ER, Stolwijk JA. Respiratory weight losses during exercise. J Appl Physiol. 1972 Apr;32(4):474-6. doi: 10.1152/jappl.1972.32.4.474. No abstract available. PMID 5026494
- [Background] Brisson GR, Boisvert P, Peronnet F, Perrault H, Boisvert D, Lafond JS. A simple and disposable sweat collector. Eur J Appl Physiol Occup Physiol. 1991;63(3-4):269-72. doi: 10.1007/BF00233860. PMID 1761019
- [Background] Buono MJ, Jechort A, Marques R, Smith C, Welch J. Comparison of infrared versus contact thermometry for measuring skin temperature during exercise in the heat. Physiol Meas. 2007 Aug;28(8):855-9. doi: 10.1088/0967-3334/28/8/008. Epub 2007 Jul 6. PMID 17664677
- [Background] Armstrong LE, Maresh CM, Gabaree CV, Hoffman JR, Kavouras SA, Kenefick RW, Castellani JW, Ahlquist LE. Thermal and circulatory responses during exercise: effects of hypohydration, dehydration, and water intake. J Appl Physiol (1985). 1997 Jun;82(6):2028-35. doi: 10.1152/jappl.1997.82.6.2028. PMID 9173973
- [Background] Temesi J, Johnson NA, Raymond J, Burdon CA, O'Connor HT. Carbohydrate ingestion during endurance exercise improves performance in adults. J Nutr. 2011 May;141(5):890-7. doi: 10.3945/jn.110.137075. Epub 2011 Mar 16. PMID 21411610
- [Background] Davis JM, Lamb DR, Burgess WA, Bartoli WP. Accumulation of deuterium oxide in body fluids after ingestion of D2O-labeled beverages. J Appl Physiol (1985). 1987 Nov;63(5):2060-6. doi: 10.1152/jappl.1987.63.5.2060. PMID 3693238